CLINICAL TRIAL: NCT06498193
Title: A Comparative Study of Cancer-related Fatigue Among Patients Receiving Home-based Palliative Care and Hospice-shared Care
Brief Title: Cancer-related Fatigue Among Patients Receiving Home-based Palliative Care
Status: Active, not recruiting | Type: Observational
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Department of Nursing, National Taipei University of Nursing and Health Sciences
Other Study IDs: 108A-07
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: to Investigate the Level of Fatigue Among Terminal Cancer Patients Receiving Home-based Hospice Care
Keywords: hospice care; cancer-related fatigue; Eastern Cooperative Oncology Group Scale

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer-related fatigue, which significantly impacts the quality of life, is prevalent among patients with terminal cancer. The experiences of fatigue, its associated needs, and the strategies for managing it are closely linked to the individual uniqueness, cultural background, and resource availability of terminal cancer patients.

DETAILED DESCRIPTION:
Fatigue is defined as any perceived or actual physical or mental tiredness that adversely affects the quality of life [7,8]. The multifaceted nature of fatigue means it manifests in various forms, including physical cognitive, and emotional. Fatigue may involve chronic exhaustion and reduced mobility that cannot be relieved by rest [9,10]. CRF is associated with cancer progression and treatment, presenting it as a painful, persistent, and subjective sensation involving physical, emotional, and cognitive tiredness or exhaustion. CRF disproportionately affects physical activities and impairs executive functions in daily life [10,11]. Factors contributing to CRF include cancer itself, treatment side effects, psychological factors such as personality traits (e.g., levels of optimism, anxiety, or depression), comorbid physical conditions, iatrogenic comorbidities, and lifestyle factors (e.g., physical activity levels) [10-12]. From the perspective of individual patients, fatigue frequently coexists with symptom clusters, such as insomnia, low mood or depression, or pain, collectively resulting in reduced daily functioning and diminished quality of life [13]. Various non-pharmaceutical interventions have demonstrated effectiveness in addressing CRF, including physical activity, mind-body approaches, and psychosocial interventions [9,14,15]. Therefore, this study aims to investigate the level of fatigue among terminal cancer patients receiving home-based hospice care, hospital-based hospice care, and hospice-shared care. The anticipated results may facilitate the enhancement of CRF management strategies

ELIGIBILITY:
Inclusion Criteria:

* (i) patients aged 20 years and above proficient in Mandarin and/or Taiwanese and willing to participate in the study; (ii) patients deemed ineligible for curative treatments by oncologists or cancer-related specialists; (iii) patients with an Eastern Cooperative Oncology Group Scale (ECOG) score of 2 or above suitable for hospice care; and (iv) patients who signed a letter of intent for hospice care,

Exclusion Criteria:

* preference on their National Health Insurance card, or signed a letter of intent for do-not-resuscitate. Patients deemed too frail

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Terminal cancer patients receiving hospital-based, hospice-shared, or home-based hospice care under the supervision of a teaching hospital in Taipei, Taiwan, were recruited through convenience sampling
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
comparing CRF scores at baseline with those after one week, | 1 week
  The BFI survey was utilized to promptly assess CRF severity and its impact on daily functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei university of nursing and health science, Taipei, Taiwan